CLINICAL TRIAL: NCT05879029
Title: Clinical Study of Jinsang Liyan Capsules Combined With Proton Pump Inhibitors in the Treatment of Laryngeal Reflux Disease (LPRD): a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Clinical Study of Jinsang Liyan Capsules Combined With PPI in the Treatment of LPRD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Xi'an Beilin Pharmaceutical Co. Ltd (Unknown)
Responsible Party: Principal Investigator, Xiang Lu, professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB20230353
Record Dates: First submitted 2023-05-08; First posted 2023-05-30 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Laryngopharyngeal Reflux
Keywords: Laryngopharyngeal Reflux; proton pump inhibitors; Jinsangliyan capsule; treatment; therapeutic evaluation
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Jinsang Liyan Capsule: oral, 0.4g/ capsule, 4 capsules, twice a day, for 8 weeks; Rabeprazole enteric-coated tablets: taken orally before breakfast, 10mg/ tablet, 2 tablets at a time, once a day, for 8 weeks;
  Interventions: Drug: Jinsang Liyan Capsule; Rabeprazole enteric-coated tablets.
- control group (Placebo Comparator): Jinsang Liyan Capsule placebo: oral, 0.4g/ capsule, 4 capsules, twice a day, for 8 weeks; Rabeprazole enteric-coated tablets: taken orally before breakfast, 10mg/ tablet, 2 tablets at a time, once a day, for 8 weeks;
  Interventions: Drug: Jinsang Liyan Capsule placebo; Rabeprazole enteric-coated tablets.

INTERVENTIONS:
Drug: Jinsang Liyan Capsule; Rabeprazole enteric-coated tablets. — Participants in the experimental group were given Jinsang Liyan Capsule + Rabeprazole enteric-coated tablets according to the requirements, and were followed up at 4 and 8 weeks. VAS and RSI scores were used to judge the improvement degree of patients' symptoms.
  Arms: experimental group
Drug: Jinsang Liyan Capsule placebo; Rabeprazole enteric-coated tablets. — Participants in the control group were given Jinsang Liyan Capsule placebo + Rabeprazole enteric-coated tablets according to the requirements, and were followed up at 4 and 8 weeks. VAS and RSI scores were used to judge the improvement degree of patients' symptoms.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of Jinsang Liyan capsule in combination with PPI versus PPI alone for the treatment of Laryngopharyngeal Reflux Disease (LPRD).

Participants will be randomly assigned in a 1:1 ratio to the experimental group or the control group. The experimental group was treated with Jinsangliyan capsule + rabeprazole enteric-coated tablets, and the control group was treated with Jinsangliyan capsule placebo + rabeprazole enteric-coated tablets. Participants were followed up at 4 weeks and 8 weeks after taking the drug to evaluate the improvement of LPRD symptoms.

Researchers will compare Experimental group and control group to see if Jinsang Liyan capsule combined with PPI treatment is superior to PPI treatment alone.

DETAILED DESCRIPTION:
According to Expert Consensus on the Diagnosis and Treatment of Throat reflux Diseases (2022, Revised edition) [J], proton pump inhibitors are the preferred drug for the medical treatment of LPRD, which can not only protect the mucosa of the upper respiratory tract and digestive tract from gastric acid damage, but also reduce the damage caused by pepsin.

At present, PPI is still the first choice for the treatment of LPRD. Other drugs include H2 blockers, gastrointestinal motonics, gastric mucosa protectors, etc. These treatments mostly focus on the response to the main pathogenic factor of stomach acid, while ignoring the symptomatic treatment of the local discomfort in the throat of LPRD patients. As a result, there are some problems in clinical treatment, such as long course of treatment, easy recurrence, easy to appear adverse reactions, poor patient compliance, etc., and it is difficult to achieve the ideal effect. Therefore, to alleviate the suffering of patients with LPRD, there is an urgent need to develop new and more effective treatments for the disease.

Many literatures have been published on the treatment of LPRD by Jinshuoliyan Pill. These studies show that Jinshuoliyan Pill has a good effect in the adjuvant treatment of laryngeal reflux disease, can significantly reduce reflux symptoms and reduce the damage to the esophageal and throat mucosa, and has certain clinical value.However, the effect of Jinsang Liyan Capsule combined with PPI in the treatment of LPRD has not been confirmed by research.

The goal of this clinical trial is to compare the efficacy of Jinsang Liyan capsule in combination with PPI versus PPI alone for the treatment of Laryngopharyngeal Reflux Disease (LPRD).

Participants will be randomly assigned in a 1:1 ratio to the experimental group or the control group. The experimental group was treated with Jinsangliyan capsule + rabeprazole enteric-coated tablets, and the control group was treated with Jinsangliyan capsule placebo + rabeprazole enteric-coated tablets. Participants were followed up at 4 weeks and 8 weeks after taking the drug to evaluate the improvement of LPRD symptoms.

Researchers will compare Experimental group and control group to see if Jinsang Liyan capsule combined with PPI treatment is superior to PPI treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* The patients who met the clinical diagnostic criteria for LPRD (by asking history and laryngoscopy, RSI score >13 or RFS score >7 points);
* No antacids or gastrointestinal motility drugs were taken within 2 weeks before enrollment.
* Be aged 18-65 years with no gender restriction;
* Patients understood and agreed to participate in this study and signed an informed consent form.

Exclusion Criteria:

* complicated with acute upper respiratory tract infection;
* combined with one of the following diseases of the digestive system: peptic ulcer, history of gastroesophageal and duodenal surgery, Zollinger-Ellison syndrome, pyloric obstruction, primary esophageal motility disorders (e.g., achalasia, scleroderma, primary esophageal spasm), drug-induced esophagitis, mycotic esophagitis, gastrointestinal malignant tumor;
* patients with severe primary diseases of heart, brain, liver, lung, kidney, blood and endocrine system, and severe psychosis without effective control;
* those who could not take medicine during pregnancy or lactation, or who were allergic to the drugs used in this study; Or unable to cooperate with medication and complete relevant records due to various circumstances;
* patients who have participated or are participating in other drug clinical trials within three months;
* patients judged by the investigator to be ineligible for trial participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
total effective rate | 2 months
  Visual analogue scale (VAS) is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
  Reflux Symptom Index (RSI) is a questionnaire that measures the severity of symptoms associated with laryngopharyngeal reflux (LPR).
  Symptom improvement rate = (VAS score before treatment - VAS score after treatment)/VAS score before treatment ×100%
  Obvious: Symptom improvement rate ≥80%; Or RSI≤13 points.
  Effective: 50% ≤ Symptom improvement rate <80%; Or RSI decreased, but still >13 points.
  Ineffective: Symptom improvement rate <50%; Or no reduction in RSI.
  Total effective rate =[(obvious + effective)/total cases]×100%

SECONDARY OUTCOMES:
RFS(reflux finding score) | 2 months
  RFS (reflux finding score) is a quantitative guide for diagnosis and treatment of laryngopharyngeal reflux. It is a score based on the presence and severity of various signs of reflux in the larynx and pharynx. The score ranges from 0 to 26, with higher scores indicating more severe reflux.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Lu, professor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Otolaryngology-Head and Neck Surgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China